CLINICAL TRIAL: NCT03220893
Title: Density MATTERS [Molecular Breast Imaging (MBI) And Tomosynthesis To Eliminate the ReServoir]
Brief Title: Molecular Breast Imaging and Digital Breast Tomosynthesis in Screening Patients With Dense Breast Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carrie Hruska, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-008522; R01CA239200 (NIH); NCI-2021-12015 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-07-15; First posted 2017-07-18 (Actual); Results first posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBT alone (Experimental): All participants undergo DBT screening
  Interventions: Procedure: Digital Breast Tomosynthesis (DBT)
- DBT + MBI (Experimental): All participants undergo DBT screening + supplemental MBI
  Interventions: Procedure: Digital Breast Tomosynthesis (DBT); Radiation: Scintimammography

INTERVENTIONS:
Procedure: Digital Breast Tomosynthesis (DBT) — DBT is standard of care breast screening
  Other Names: DBT; Digital Breast Tomosynthesis; Digital Tomosynthesis Mammography; Digital Tomosynthesis of the Breast
Radiation: Scintimammography — Undergo MBI
  Other Names: Breast-Specific Gamma Imaging; MBI; Miraluma Scan; Miraluma Test; Molecular Breast Imaging; Nuclear Medicine Breast Imaging; sestamibi breast imaging; Sestamibi Scintimammography
  Arms: DBT + MBI

SUMMARY:
This study compares molecular breast imaging (MBI) and digital breast tomosynthesis (DBT) in screening patients with dense breast tissue. Breast imaging may help doctors find breast cancer sooner, when it may be easier to treat. Molecular breast imaging (MBI) uses an injection of a small amount of radioactive material that is taken up in tissues of the body that are actively changing, such as breast cancer. A specialized camera, called a gamma camera, takes pictures of the gamma rays emitted by this material. MBI may detect cancers that are not visible on mammograms. This study may help researchers determine how MBI testing compares to DBT screening.

DETAILED DESCRIPTION:
This study includes women age 40-75 who are presenting for breast cancer screening and had mammographically dense breasts on their last mammogram. Participants undergo annual DBT and MBI screening for two years. The primary aim for this study is to compare the rate of detection of invasive cancers between DBT alone vs. the combination of DBT with supplemental MBI at the first year of screening.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a consenting female age 40-75 years
* Patient is scheduled for routine screening DBT
* Patient is asymptomatic for breast disease
* Patient had heterogeneously dense or extremely dense breasts on most recent prior mammography examination (Breast Imaging Reporting and Data System [BI-RADS] c or d) within 24 months of enrollment
* Patient is able to participate fully in all aspects of the study (completing study visits and study data collection)
* Patient understands and signs the study informed consent
* Patient anticipates being able to return one year after study enrollment to complete the second round of screening

Exclusion Criteria:

* Patient is currently pregnant or plans to become pregnant during the course of the study
* Patient is currently lactating
* Patient has had a prior MBI
* Patient has had a prior whole breast ultrasound (WBUS) for screening, with either a hand-held ultrasound probe or automated system, within 12 months prior to study enrollment
* Patient has had a prior breast MRI
* Patient has had a prior contrast-enhanced mammogram (contrast enhanced spectral mammography [CESM] or contrast-enhanced digital mammography [CEDM])
* Patient is concurrently participating in any other breast imaging research studies that involve undergoing additional breast imaging tests beyond routine screening with mammography, including but not limited to contrast-enhanced mammography, WBUS, MBI, or contrast-enhanced breast MRI
* Patient has had a breast biopsy within 3 months prior to study enrollment
* Patient has had breast surgery within 12 months prior to study enrollment
* Patient is currently undergoing treatment for breast cancer or planning surgery for a high-risk breast lesion (atypical ductal hyperplasia [ADH], atypical lobular hyperplasia [ALH], lobular carcinoma in situ [LCIS], papilloma, radial scar)
* Patient is currently taking a chemoprevention agent for breast cancer risk reduction or osteoporosis prevention (tamoxifen, raloxifene, anastrazole, letrozole, exemestane)
* Patient has a known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder study adherence

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3023 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie B. Hruska, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (5):
- United States (5):
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - M D Anderson Cancer Center, Houston, Texas
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred from June 2017 to July 2022 through consecutive sampling.
Groups:
- All Participants: All participants are screened with DBT and MBI
Period: DBT Alone
Arm/Group | All Participants
Started | 2978
Completed | 2978
Not Completed | 0
Period: DBT + MBI
Arm/Group | All Participants
Started | 2978
Completed | 2978
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 2978 participants met eligibility criteria and had both DBT and MBI screening performed
Arm/Group | All Participants
Number analyzed (Participants) | 2978
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2978
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7
  Asian | 59
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 268
  White | 2592
  More than one race | 4
  Unknown or Not Reported | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 77
  Not Hispanic or Latino | 2833
  Unknown or Not Reported | 68

OUTCOME MEASURES:

1. Primary Outcome: Rate of Detection of Invasive Cancers
Description: Compare the rate of detection of invasive cancers between DBT alone versus (vs.) the combination of digital breast tomosynthesis (DBT) with supplemental molecular breast imaging (MBI) at initial (year 1) screening. For each modality, the detection rate of invasive cancers will be estimated as the proportion of participants in the analysis set who had an invasive cancer detected by the modality and verified by pathology.
Time Frame: At year 1 screening
Population: Of 2978 participants screened with DBT alone and with DBT + supplemental MBI, 23 participants had invasive breast cancer detected.
Measure: Count of Participants; unit: Participants
Groups:
- Observational (MBI, DBT): Participants undergo DBT and MBI at year 0 and year 1 screening.
Arm/Group | Observational (MBI, DBT)
Number analyzed (Participants) | 23
Participants
  Invasive cancers detected by DBT alone | 9
  Additional invasive cancers detected by supplemental MBI | 14

ADVERSE EVENTS:
Time Frame: 365 days after screening
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/2978
Serious Adverse Events (participants affected / at risk) | 0/2978
Other Adverse Events (participants affected / at risk) | 0/2978

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT03220893/Prot_SAP_000.pdf